CLINICAL TRIAL: NCT00444288
Title: PCOS Twin Study - Environmental Factors in the Development of Polycystic Ovary Syndrome, Phase 2
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907112; 07-E-N112
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-03-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Cystic Ovaries; Hyperandrogenism; Anovulation; Concordance Rates; Baseline Heritability; Polycystic Ovary Syndrome; POS
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Cysts; Hyperandrogenism; Anovulation

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Polycystic Ovary Syndrome, or PCOS, is the most common endocrine disorder in women. Depending on the strictness of the diagnostic criteria used, it is thought to occur in about 6-10% of all women, many of whom do not know they have the syndrome. Women with PCOS produce abnormally high levels of male hormones (hyperandrogenism); this counteracts their ovaries' ability to make enough of the female hormones estrogen and progesterone needed for normal menstruation. PCOS is the number one cause of hormonally related infertility and also increases women's risks for diabetes, high blood pressure, hypercholesteremia, cardiovascular disease and certain cancers. It is currently unclear to what extent PCOS and PCOS-associated traits (hyperandrogenisms, hyperinsulinemia, insulin resistance, type 2 diabetes, dyslipidemia, hypertension, obesity, and coronary artery disease) are the results of environmental factors or genetic predisposition. Therefore, the NIEHS Program in Clinical Research is conducting a multi-phase twin study to measure the extent of PCOS heritability and to identify environmental and genetic factors involved in the development of PCOS. The proposal described here is for Phase 2 of this study. The goals of Phase 2 are to: 1) establish more reliable concordance rates and baseline heritability estimates for PCOS in MZ and DZ twins; and 2) establish a cohort of intact MZ and DZ female twin pairs as a resource for future studies.

In Phase 1, about 1500 individual female twins were identified from the Mid-Atlantic Twin Registry (MATR) based on self report of a history of irregular periods and/or cystic ovaries in the MATR General Health Screening Questionnaire. Those twins were surveyed by phone for other traits associated with PCOS. In Phase 2, the twins most likely to have PCOS based on their answers to the Phase 1 phone survey will be recontacted for further PCOS screening. This includes providing a blood sample for measuring bioavailable testosterone (BaT) levels. Women with elevated BaT levels are likely to have PCOS. The women with elevated levels will then be asked to undergo a medical evaluation for PCOS confirmation. This includes a physical exam, medical history, ultrasound, 2-hour glucose tolerance and other biochemical blood tests, and a Ferriman-Gallwey evaluation for abnormal hirsutism (another characteristic of PCOS). The women will also be tested for pregnancy and zygosity. Their female co-twins will be invited to undergo...

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome, or PCOS, is the most common endocrine disorder in women. Depending on the strictness of the diagnostic criteria used, it is thought to occur in about 6-10% of all women, many of whom do not know they have the syndrome. Women with PCOS produce abnormally high levels of male hormones (hyperandrogenism); this counteracts their ovaries' ability to make enough of the female hormones estrogen and progesterone needed for normal menstruation. PCOS is the number one cause of hormonally related infertility and also increases women's risks for diabetes, high blood pressure, hypercholesteremia, cardiovascular disease and certain cancers. It is currently unclear to what extent PCOS and PCOS-associated traits (hyperandrogenism, hyperinsulinemia, insulin resistance, type 2 diabetes, dyslipidemia, hypertension, obesity, and coronary artery disease) are the results of environmental factors or genetic predisposition. Therefore, the NIEHS Program in Clinical Research is conducting a multi-phase twin study to measure the extent of PCOS heritability and to identify environmental and genetic factors involved in the development of PCOS. The proposal described here is for Phase 2 of this study. The goals of Phase 2 are to: 1) establish more reliable concordance rates and baseline heritability estimates for PCOS in MZ and DZ twins; and 2) establish a cohort of intact MZ and DZ female twin pairs with PCOS as a resource for future studies.

In Phase 1, about 1500 individual female twins were identified from the Mid-Atlantic Twin Registry (MATR) based on self report of a history of irregular periods and/or cystic ovaries in the MATR General Health Screening Questionnaire. Those twins were surveyed by phone for other traits associated with PCOS. In Phase 2, the twins most likely to have PCOS based on their answers to the Phase 1 phone survey will be recontacted for further PCOS screening. One or both twins in a pair will be screened for elevated levels of testosterone (total and free testosterone, bioavailable testosterone or BaT; free androgen index or FAI). Hyperandrogenism is one of the hallmark traits of PCOS and can be exhibited either biochemically (elevated testosterone) or clinically (hirsutism, acne, hair loss, alopecia, other). If one twin in a pair has an elevated BaT level, then both twins in the pair will be asked to undergo a medical evaluation for PCOS confirmation. This includes a physical exam, medical history, ultrasound, 2-hour glucose tolerance and other biochemical blood tests, and a Ferriman-Gallwey evaluation for abnormal hirsutism (another characteristic of PCOS). The women will also be tested for pregnancy and zygosity. Their female co-twins will be invited to undergo a similar medical evaluation.

Depending on their PCOS traits, twin pairs in which neither member has elevated testosterone levels might be asked to undergo the medical evaluation as well. In clinical practice, PCOS diagnoses are often made on women with normal testosterone levels if they have other certain PCOS traits. The determination to include pairs in which both members have normal testosterone levels will be made depending on their collective PCOS traits that they reported on their Phase 1 survey.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be included in this study, primary twins must:

1. Be a premenopausal female twin over the age 18 (this will be asked during recruitment).
2. Have a living female co-twin (this will be asked during recruitment).
3. Have a history of probable PCOS defined by having one or more of the following criteria as self-reported in the Phase 1 PCOS survey. These traits will be confirmed during medical evaluation:

   1. History of chronically irregular menstrual cycles
   2. History of hirsutism
   3. History of hair loss
   4. Cysts in ovaries
   5. Body-mass index greater than 25
   6. Acne
4. Be able and willing to give informed consent.
5. Agree to undergo a medical evaluation for PCOS.

To be included in this study, co-twins must:

1. Be a premenopausal female twin over the age of 18 (this will be asked during recruitment).
2. Be able and willing to give informed consent.
3. Agree to undergo a medical evaluation for PCOS.

EXCLUSION CRITERIA:

Women will be excluded from the study if they are pregnant or have given birth within the past six months.

Women will also be excluded if they are currently menopausal or past menopause.

Women with any condition that, in the opinion of the investigators, could affect the validity of the study results will be excluded from participating.

Subjects will not be excluded based on race, ethnicity or religion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-02-27; Study Completion 2010-03-01

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States